CLINICAL TRIAL: NCT04462939
Title: Effects of Multiple Micronutrients, Lutein and Docosahexaenoic Acid (DHA) Supplementation During Lactation on Human Milk Nutrient Content, Maternal Blood Biomarkers and Infant Anthropometric Parameters
Brief Title: Study to Learn About the Effect of Elevit (a Food Supplement Containing Several Vitamins, Minerals, Lutein and DHA) on the Nutrient Content in the Breast Milk and Blood of Women During Breastfeeding Period and on Babies' Physical Growth Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18737
Record Dates: First submitted 2020-05-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Healthy Lactating Mother
MeSH Terms: interventions — Postnatal Care; Lutein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy lactating women - Supplement (Experimental): At randomization (Visit 2), from four to six weeks after delivery, eligible actating women will be equally randomized to one of the study arms (supplementation arm or placebo arm) and will assume the supplement or placebo once daily for a duration of 12 weeks.
  Interventions: Dietary Supplement: Elevit Breastfeeding & Postnatal Care
- Healthy lactating women - Placebo (Placebo Comparator): At randomization (Visit 2), from four to six weeks after delivery, eligible actating women will be equally randomized to one of the study arms (supplementation arm or placebo arm) and will assume the supplement or placebo once daily for a duration of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Elevit Breastfeeding & Postnatal Care — Multi-micronutrients, lutein and DHA soft gel capsules; one capsule daily, oral
  Other Names: BAY987816 - Multi-micronutrients, lutein & DHA
  Arms: Healthy lactating women - Supplement
Drug: Placebo — No active ingredients except of 225 μg iodine; One capsule daily, oral
  Arms: Healthy lactating women - Placebo

SUMMARY:
The aim of the study is to learn about the effect of multi-micronutrient, lutein and DHA supplementation (Elevit Breastfeeding & Postnatal Care) on the breast milk nutrient composition and babies physical growth parameters.

Mothers participating in this study received either Elevit or placebo orally once a day for 12 weeks starting from 4 to 6 weeks after delivery. Blood, urine and milk samples were collected from the mothers and physical parameters like size and weight were collected from the babies to assess the effect of the supplementation.

ELIGIBILITY:
Inclusion Criteria for women:

* Healthy pregnant women aged 18 to 45 years (inclusive) in their third trimester of pregnancy who are expected to give birth to a healthy single full-term infant;
* Hb > 105 g/L;
* Intention to breastfeed for at least four months (no more than one bottle or 10% of total milk intake daily as formula);
* Omnivorous diet;
* Not intent to take multivitamin supplements, DHA supplements, lutein supplements or any combination of the aforementioned after giving birth except for iodine and iron;
* Seronegative for Human Immunodeficiency Virus (HIV), Hepatitis B, and Hepatitis C at screening;
* Pregnant women who, in the opinion of the Investigator, are willing and able to participate in all scheduled visits, to adhere to the study plan, to laboratory tests and to all other study related procedures according to the clinical protocol;
* Pregnant women providing a personally signed and dated informed consent willing to participate in the study and to adhere to all study procedures including the assessments done to the infant, indicating that they have been informed of all pertinent aspects of the trial and that they understood and accepted these, prior to admission to the study.

Inclusion Criteria for infants:

* Full term/gestational age > 37 weeks < 43 weeks and birth weight adequate for gestational age;
* Apgar score at 5 minutes after birth > 7;
* No indication of abnormal neurodevelopment.

Exclusion Criteria for women:

* Physical (including vital signs e.g. blood pressure, pulse rate), hematological and clinical-chemical parameters deviating from normal and with clinical relevance in the opinion of the investigator;
* Any serious infection (acute or chronic) at screening and randomization;
* Any history of or current metabolic diseases (e.g. diabetes, hypothyroidism, and other metabolic diseases);
* Less than 12 months from previous delivery;
* Any history of or current diseases, which are associated with malabsorption, or other severe diseases of the gastrointestinal tract (e.g. chronic inflammatory bowel disease, iron accumulation, iron utilization disorders);
* Any history of or current neurological, cardiac, endocrine or bleeding disorders;
* Specific diets (e.g. vegan, vegetarian, celiac);
* Pre-pregnancy body mass index (BMI) < 18.5 or > 30 kg/m2;
* Diagnosed or suspected malignant or premalignant disease;
* Current clinically significant depression;
* Not willing, or unable for medical reasons to interrupt any intake of pharmaceuticals or dietary supplements which may interact with any of the ingredients of the trial product (i.e. fluoroquinolones, bisphosphonates, levodopa, levothyroxine, penicillamine, antibiotics containing tetracycline or trietine) during the study supplementation period (From Visit 2 (Randomization) until Visit 4 (EoS));
* History of or current diseases where vitamin, mineral, trace element, lutein or DHA supplementation might be not recommended / contraindicated (such as sickle cell anemia, copper metabolism disorders (Wilson's disease), renal disease, nephrolithiasis, urolithiasis, hypercalcemia, hypercalciuria, hepatobiliary diseases, existing hypervitaminosis, iron metabolism disorders, hypermagnesemia);
* Any pregnancy complications or adverse pregnancy outcomes in current pregnancy that may affect micronutrient metabolism or status (e.g. preeclampsia, eclampsia, polyhydramniosis, placental insufficiency);
* Diagnosed congenital abnormalities in current pregnancy;
* Current smoker or smoker during current pregnancy.

Main exclusion criteria for infants:

* Congenital anomalies;
* Obvious gastrointestinal or metabolic disorders;
* Perinatal hypoxia;
* Preterm birth;
* Very low birth weight (VLBW).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in human milk total lipid docosahexaenoic acid (DHA) content: % DHA concentration relative to total milk | At Baseline and 6 weeks and 12 weeks
  The primary endpoint will be analyzed using the analysis of covariance (ANCOVA) with supplementation as fixed effect and baseline value as covariate.

SECONDARY OUTCOMES:
Change from baseline in blood parameters: % concentration relative to total milk | At Baseline and 6 weeks and 12 weeks
  Fatty acids (FA) in plasma and glycerophospholipids (GPL); DHA/total fatty acid (TFA) ratio; IFN-gamma; TGF-beta; Folic acid, Vitamin B12 and homocystein; 25-Hydroxivitamin D; Alpha-tocopherol and retinol; Carotenoids (lutein, zeaxanthin, beta-cryptoxanthin, lycopene, carotene)
Change from baseline in milk parameters: % concentration relative to total milk | At Baseline and 6 weeks and 12 weeks
  Total lipids; DHA/total FA ratio; Milk macronutrient content; IFN-gamma; TGF-beta; Alpha-tocopherol and retinol; Carotenoids (lutein, zeaxanthin, beta-cryptoxanthin, lycopene, carotene)
Change from baseline: maternal height | At Baseline and 12 weeks
Change from baseline: maternal weight | At Baseline and 12 weeks
Change from baseline: Maternal BMI kg/m2 | At Baseline and 12 weeks
Change from baseline: Maternal fatigue questionnaire | At Baseline and 6 weeks and 12 weeks
Change from baseline: Maternal food frequancy questionnaire | At Baseline and 6 weeks and 12 weeks
Change from baseline: Infant weight | At Baseline and 6 weeks and 12 weeks
Change from baseline: Infant length | At Baseline and 6 weeks and 12 weeks
Change from baseline: Infant Calculation of Weight Standard Deviation Scores (SDS) | At Baseline and 6 weeks and 12 weeks
Change from baseline: Infant Calculation of Length Standard Deviation Scores (SDS) | At Baseline and 6 weeks and 12 weeks
Number of Adverse Events (AEs) | Up to 13 weeks
Severity of AEs | Up to 13 weeks
AE relationship to the investigational product | Up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Germany (3):
  - Gynäkologische Gemeinschaftspraxis Freising, Freising, Bavaria
  - Praxis Hr. E. Goeckeler-Leopold, Geseke, North Rhine-Westphalia
  - Praxis Fr. Dr. K. Maar, Berlin